CLINICAL TRIAL: NCT06048549
Title: Effect Of Obesity on The Outcome Of Mechanically Ventilated Chronic Obstructive Pulmonary Disease Patients
Brief Title: The Effect of Obesity in COPD Mechanically Ventilated Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Asmaa Gamal Abd Elhamied, Assistant lecturer at Assiut university hospital, Assiut University
Other Study IDs: Obesity COPD Patients
Record Dates: First submitted 2023-09-16; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Effects of Obesity on COPD Mechanically Ventilated Patients

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Study the relationship between the body mass index and duration of mechanical ventilation & complications in mechanically ventilated COPD patients.

Study the effect of obesity on mortality rate of COPD mechanically ventilated patients.

Determine prevalence of obesity in mechanically ventilated COPD patients.

DETAILED DESCRIPTION:
Obesity has become a global epidemic with prevalence rising both in developed and developing countries. The percentage of patients with obesity in the intensive care unit (ICU) can be expected to increase concomitantly or even more since obesity increases the risk for a more severe disease course with more need for ICU admission and mechanical ventilation .

Obesity, especially abdominal obesity (android fat distribution) and severe obesity, results in altered respiratory anatomy and physiology and, therefore, complicated airway management and adapted ventilator settings during mechanical ventilation. Obesity appears to be associated with an increased risk of acute respiratory distress syndrome (ARDS) and infection, mainly pneumonia probably related to an imbalanced production of adipokines. In ventilated patients, obesity increases ICU length of stay and the duration of mechanical ventilation .

Obesity is relatively common among individuals with COPD, corresponding to 20%-35% of patients with COPD. Increasing evidence suggests that obesity is a risk factor for impaired quality of life, exercise intolerance, and suboptimal disease control in COPD .

ELIGIBILITY:
Inclusion Criteria:

* Adult patients of both genders more than 18 years old admitted at RICU, diagnosed COPD and need mechanical ventilation from August 2023 to August 2024.

Exclusion Criteria:

patients less than 18 years old. patients who refused to participate in the research. patients with missing data.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients of both genders more than 18 years old admitted at RICU, diagnosed COPD and need mechanical ventilation from August 2023 to August 2024.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-10 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Study the effect of obesity on morbidity and mortality rate of COPD mechanically ventilated patients. | one year
  Study the relationship between the body mass index and duration of mechanical ventilation & complications in mechanically ventilated COPD patients.

IPD SHARING:
Plan to Share IPD: No